CLINICAL TRIAL: NCT02490683
Title: The Effect of Soy-based Dietary Supplements on Cardiometabolic Risk Factors in Individuals at High Risk for Cardiovascular Disease
Brief Title: Effects of Soy Based Dietary Supplements on Cardiometabolic Risk Factors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, DrPH, MD, Loma Linda University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 5150056
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Cardiovascular Risk Factors
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Luna Rich X (Experimental): Luna Rich X©: 500 mg/ day in 4 pills of lunasin-enriched soy protein concentrate Reliv Now: 19 grams of powder/day, that subject will mix and consume daily with water or a beverage they commonly drink
  Interventions: Dietary Supplement: Luna Rich X
- Reliv Now (Experimental): 19 grams of power/day, that subjects will mix and consume daily with water or a beverage they commonly drink
  Interventions: Dietary Supplement: Reliv Now
- Placebo (Placebo Comparator): Placebo pills containing starch (provided by Reliv International, Inc.)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Luna Rich X
  Arms: Luna Rich X
Dietary Supplement: Placebo — Starch pill/or powder manufactured to mimic Luna Rich X and Reliv Now
  Arms: Placebo
Dietary Supplement: Reliv Now
  Arms: Reliv Now

SUMMARY:
This study will test the effect of both Luna Rich X© and Reliv Now© against placebo pills or powder (control) on blood lipids. It will also explore the potential effects of these dietary supplements on inflammation markers and other biological and anthropometric measures. The study intervention will be 30 weeks in length. Twenty four subjects with 2 or more cardiometabolic risk factors will be randomized to participate in the study.

DETAILED DESCRIPTION:
Primary Objective To test the effects of Luna Rich X©, and Reliv Now© on serum lipids and selected inflammatory and oxidative parameters.

Secondary Objective To explore the potential effects of Luna Rich X© and Reliv Now© on body weight and adiposity.

Hypotheses

1. Eight-week supplementation of formulated lunasin-enriched soy concentrate (Luna Rich X©) in adults at risk for cardiovascular disease will improve their serum lipid profile and reduce inflammatory parameters.
2. Eight-week supplementation of a formulated soy-based powder (Reliv Now) plus Luna Rich X in adults at risk for cardiovascular disease will improve their serum lipid profile and reduce inflammatory parameters.

Study Protocol

Recruitment of Subjects Subjects will be recruited from out-patient clinics in or near Loma Linda University. In collaboration with the medical personnel of the Family and Internal Medicine clinics of the Loma Linda University and Beaver Medical Group, interested clients/patients will be referred to the study. Potential subjects will be informed about the study by the physician, nurse or other clinic personnel and will be given a flyer. Individuals will make their own decision whether or not to participate in the study. The clients/patients who will be interested in participating in the study will contact the investigators via the provided phone numbers. A dedicated telephone line and webpage will provide both additional information to interested individuals and a means to screen out subjects by the study personnel. Potential subjects will first be screened by study personnel, and then directed to a clinical laboratory at Loma Linda University for determination of biochemical parameters on which the eligibility for the study will be determined.

Dietary Interventions

* Luna Rich X©: 500 mg/ day in 4 pills of lunasin-enriched soy protein concentrate
* Reliv Now: 19 grams of powder/day, that subject will mix and consume daily with water or a beverage they commonly drink.
* Control: Placebo pills containing starch (provided by Reliv International, Inc.)

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 35-75 years of age, at high risk for cardiovascular disease, i.e. with 2 or more risk factors:

* Present tobacco smoker
* Arterial hypertension (BP ≥140/90 mm Hg or treatment)
* LDL-cholesterol ≥130 mg/dl
* HDL-cholesterol ≤ 40 mg/dl
* Triglycerides ≥150 mg/dl
* Fasting blood glucose ≥110 mg/dl
* Overweight or obesity (BMI ≥ 25 kg/m2)
* Family history of premature heart disease

Exclusion Criteria:

1. Uncontrolled renal/hepatic/endocrine disease
2. Abnormal blood chemistry profile
3. Familial hypercholesterolemia or other genetic dyslipidaemia
4. Intake of lipid-lowering drugs and dietary products including plant sterols/stanols
5. High Framingham risk or medical condition in which statin therapy is considered necessary by a treating physician
6. Hypersensitive or allergic to soy
7. Alcohol or drug addiction/abuse
8. Diabetics
9. Impossibility or lack of interest to follow the dietary intervention

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Serum Lipid profile | baseline- 30 weeks
  Serum Low density cholesterol, high density cholesterol, apo Lipoprotein A and B, apo E allele genetic typing and triglycerides will be measured from the by performing lab tests.
Inflammatory and oxidative parameters | baseline- 30 weeks
  hs-CRP (highly sensitive C-reactive protein), TNF-alpha (tissue necrosis factor alpha), IL-6 (Interleukin 6), ox-LDL (oxidized low density lipoprotein), TBARS (thiobarbituric acid reactive substances) lipid peroxides, 8-OHdG (8-hydroxy-2-deoxyguanosine) will be measured via lab tests

SECONDARY OUTCOMES:
Hormones | baseline- 30 weeks
  : adiponectin, leptin, insulin, C-peptide (C-peptide of insulin); and fasting glucose and hemoglobin A1c. will be measured via lab tests
Compliance | baseline -30 weeks
  , blood samples will be taken for testing levels of lunasin and/or its metabolites as biological marker(s) of the treatment compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabate, DrPH, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University School of Public Health, Loma Linda, California, United States